CLINICAL TRIAL: NCT05878470
Title: Reducing Self-stigma Using Brief Video Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Doron Amsalem, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8432
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Stigma, Social; Mental Health Disorder
MeSH Terms: conditions — Social Stigma; Mental Disorders | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief video intervention (Experimental): Brief (119 seconds) social contact-based video
  Interventions: Behavioral: video
- Non-intervention control (No Intervention): Non-intervention control

INTERVENTIONS:
Behavioral: video — A brief (119 seconds) social contact-based video. The video presented a young Black man in his early twenties, a professional actor, sharing his scripted personal story of struggles with psychotic illness and raising themes of recovery and hope.
  Arms: Brief video intervention

SUMMARY:
Stigma is a profound obstacle to care. Self-stigma decreases sense of self-competency, as well as healthcare seeking and treatment adherence and creates barriers to pursuing employment, independent living, and fulfilling social life. For example, people with mental disorders avoid, delay, or drop out of treatment due to a fear of labeling and discrimination or experience treatments as ineffective or disrespectful. Therefore, reducing self stigma can reduce self-blame, improve self-confidence and provide support for people living with mental illness.

In a prior study, the investigators developed a short video intervention to reduce self-stigma among people with schizophrenia. The investigators would like to test the efficacy of this video using Prolific (a crowdsourcing platform). Specifically, the investigators are interested in recruiting 1,200 Prolific participants, ages 18-35, who mentioned in their profile while enrolling to Prolific that they have a mental health condition, and randomized them into watching the newly developed video to reduce self-stigma or participate in the non-intervention control arm. Participants will be invited to participate in a follow-up survey 30 days after completing the first survey.

DETAILED DESCRIPTION:
The primary objective of this study is to test the video efficacy in reducing self stigma among 1,200 Prolific users who mentioned in their profile while enrolling to Prolific that they have a mental health condition (600 in an intervention group, and 600 in a non-intervention control group). The study participants will be invited to participate in a 30-day follow up questionnaire. The investigators hypothesize finding a reduced level of self-stigma among those who watch the intervention video.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18-35-year-old
* US residents
* Those who answered yes to "Do you have or have you had a diagnosed, ongoing mental health/illness/condition?"

Exclusion Criteria:

* Non English-speaking
* Non US residents
* Age younger than 18 or older than 35
* People who replied no to the question on ongoing mental health

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1214 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Self-stigma | Baseline
  The investigators assessed self-stigma using 23 items across six domains: Stereotype Endorsement, Alienation, Stigma Resistance, Perceived Devaluation Discrimination, Secrecy, and Recovery Assessment Scale.
Self-stigma | Post (immediately after the intervention and for the control immediately after doing the baseline survey)
  The investigators assessed self-stigma using 23 items across six domains: Stereotype Endorsement, Alienation, Stigma Resistance, Perceived Devaluation Discrimination, Secrecy, and Recovery Assessment Scale.
Self-stigma | 30 day follow up
  The investigators assessed self-stigma using 23 items across six domains: Stereotype Endorsement, Alienation, Stigma Resistance, Perceived Devaluation Discrimination, Secrecy, and Recovery Assessment Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amsalem D, Jankowski SE, Yanos P, Yang LH, Markowitz JC, Rogers RT, Stroup TS, Dixon LB, Pope LG. Randomized Controlled Trial of a Brief Video Intervention to Reduce Self-Stigma of Mental Illness. J Clin Psychiatry. 2024 Mar 6;85(1):23m15034. doi: 10.4088/JCP.23m15034. PMID 38451170